CLINICAL TRIAL: NCT01728883
Title: Evaluation of New Self-Test Visual Function Assessment System for Diabetic Retinopathy
Brief Title: Diabetic Retinopathy And the Myvisiontrack® (DRAMA) Study
Acronym: DRAMA
Status: Completed | Type: Observational
Sponsor: Vital Art and Science Incorporated (Industry)
Collaborators: National Eye Institute (NEI) (NIH); Retina Foundation of the Southwest (Other); University of Texas Southwestern Medical Center (Other); Texas Retina Associates (Other)
Responsible Party: Sponsor
Other Study IDs: 2R44EY020016-03 (NIH); 2R44EY020016 (NIH)
Record Dates: First submitted 2012-11-13; First posted 2012-11-20 (Estimated); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: Diabetic Retinopathy; Diabetic Macular Edema
Keywords: Diabetic Retinopathy; Diabetic Macular Edema; Macular Edema; Maculopathy; home monitoring; shape discrimination hyperacuity; Psychophysical Testing
MeSH Terms: conditions — Diabetic Retinopathy; Macular Edema; Macular Degeneration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Diagnosed DR/DME requiring treatment: Patients diagnosed as diabetic retinopathy(DR) and/or diabetic macular edema (DME) and requiring treatment at the time they are recruited into the Study. Patients will be home vision monitoring using myVisionTrack®.
  Interventions: Device: Home vision monitoring using myVisionTrack®

INTERVENTIONS:
Device: Home vision monitoring using myVisionTrack® — Patients will be asked to test their vision at home twice per week using myVisionTrack® during the study period.
  Other Names: myVisionTrack® Model 0004

SUMMARY:
The purpose of this study is to determine the effect of enhancements to the myVisionTrack® in regards to patient compliance and test-retest variability. Additionally, the ability of myVisionTrack® to detect changes in vision function will be evaluated.

DETAILED DESCRIPTION:
The results of this study will provide the basis for patient self-monitoring of visual function with the myVisionTrack®, and for reporting, storage, and maintenance of collected data. The myVisionTrack® is intended to be used remotely by patients to monitor their disease. In the case of significant changes, patients will be prompted to visit their ophthalmologist. It is hypothesized that this can lead to earlier detection of disease progression, which, in turn, can lead to earlier treatment and better prevention against vision loss due to diabetic retinopathy (DR).

ELIGIBILITY:
Inclusion Criteria:

* DR or AMD requiring treatment at time of study initiation
* Macular edema involving the central subfield based on clinical judgment
* No noticeable central subfield atrophy
* Patients willing and able to comply with all study and follow-up procedures (including the handling of the myVisionTrack™ device)

Exclusion Criteria:

* Any ocular pathology other than DR or AMD
* Any other concurrent systemic illness affecting the retina and visual function
* Dementia or other neurological or psychological limitation that would prevent patients from performing self-testing of visual function
* Past (within the prior 6 months) or current use of, or likely need for, systemic medications that are known to be toxic to the lens, retina, or optic nerve
* Use of investigational drugs at the time of screening, or within 60 days (excluding vitamins and minerals)
* Pregnancy

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diabetic retinopathy requiring treatment
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2013-04; Primary Completion 2016-04 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Test efficacy of the test algorithm improvements | Twelve months
  To test the efficacy of test algorithm improvements and usability enhancements on the overall rate of patient compliance and on test-retest variability.

SECONDARY OUTCOMES:
Refine the decision rule | Twelve months
  To refine the decision rule so as to select optimal cutoff values to achieve desired sensitivity and specificity of self-test
Can improved testing algorithm minimize test time? | Twelve months
  To determine if the improved testing algorithm can minimize the length of testing while maintaining or improving accuracy
Assess patient satisfaction with the test | Twelve months
  To assess patient satisfaction regarding the use of myVisionTrack™

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Zhong Wang, PhD, Study Chair — Retina Foundation of the Southwest
Locations (2):
- United States (2):
  - Retina Foundation of the Southwest, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
DME Monitoring Results presented at ARVO on May 2, 2016. Additional results planned.